CLINICAL TRIAL: NCT00001526
Title: Trial of Treatment of Non-Infectious Intermediate and Posterior Uveitis With Humanized Anti-Tac Antibody Therapy
Brief Title: ANTI-TAC THERAPY FOR UVEITIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960096; 96-EI-0096
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Uveitis
Keywords: Uveitis; Interleukin 2 Receptor; Daclizumab; HAT; Zenapax; Interleukin 2
MeSH Terms: conditions — Uveitis; Diabetes Mellitus, Insulin-Dependent, 10 | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab (Zenapax)

SUMMARY:
Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects. Consequently, an effective treatment with a safer side effect profile is highly desirable.

This pilot study has permitted enrollment of up to 12 adults with non-infectious intermediate or posterior uveitis who require treatments to maintain visual function. This extended protocol began with an evaluation of the safety and potential efficacy of intravenous (IV) daclizumab treatments for uveitis while reducing or eliminating standard medications commensurate with the standard of care. As subcutaneous (SC) daclizumab treatments become available, eligible participants will be offered continuing daclizumab treatments using the new SC formulation, though they may elect to remain on the IV treatments. If the therapeutic benefit is sustained using the SC formulation, maintenance therapy will continue as clinically indicated. Participants who repeatedly fail the SC therapy will be permitted to revert to the IV daclizumab regimen they previously used, or may exit the study as treatment failures. SC treatments begin with a short SC induction at 2 mg/kg followed by 1 mg/kg treatments on a 4-week schedule as the protocol originally specified. Participants will be monitored routinely when each dose is received and additionally will participate in pharmacokinetic studies to monitor SC formulation bioavailability.

Daclizumab is a humanized anti-Tac monoclonal antibody (HAT, Zenapax) that interferes with inflammatory processes by its involvement with the interleukin 2 receptor (IL-2R). During the first 5 years of this study, only an IV product was available. The SC formulation is now available containing the same daclizumab drug product. Preliminary studies indicate that the SC formulation is well tolerated by normal control subjects and other autoimmune disease patients at repeated doses up to 2 mg/kg.

The primary objectives are to examine the safety and potential efficacy of IV and later, SC daclizumab, while continuing to reduce other immunosuppressive medications commensurate with the standard of care. Primary safety outcomes are the discontinuation of study therapy due to reduced vision or the occurrence of adverse events. Secondary outcome measures include visual acuity and the grading of immunosuppressive medications, anterior chamber and vitreous cells, and vitreous haze.

DETAILED DESCRIPTION:
Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects. Consequently, an effective treatment with a safer side effect profile is highly desirable.

This pilot study has permitted enrollment of up to 12 adults with non-infectious intermediate or posterior uveitis who require treatments to maintain visual function. This extended protocol began with an evaluation of the safety and potential efficacy of intravenous (IV) daclizumab treatments for uveitis while reducing or eliminating standard medications commensurate with the standard of care. As subcutaneous (SC) daclizumab treatments become available, eligible participants will be offered continuing daclizumab treatments using the new SC formulation, though they may elect to remain on the IV treatments. If the therapeutic benefit is sustained using the SC formulation, maintenance therapy will continue as clinically indicated. Participants who repeatedly fail the SC therapy will be permitted to revert to the IV daclizumab regimen they previously used, or may exit the study as treatment failures. SC treatments begin with a short SC induction at 2 mg/kg followed by 1 mg/kg treatments on a 4-week schedule as the protocol originally specified. Participants will be monitored routinely when each dose is received and additionally will participate in pharmacokinetic studies to monitor SC formulation bioavailability.

Daclizumab is a humanized anti-Tac monoclonal antibody (HAT, Zenapax) that interferes with inflammatory processes by its involvement with the interleukin 2 receptor (IL-2R). During the first 5 years of this study, only an IV product was available. The SC formulation is now available containing the same daclizumab drug product. Preliminary studies indicate that the SC formulation is well tolerated by normal control subjects and other autoimmune disease patients at repeated doses up to 2 mg/kg.

The primary objectives are to examine the safety and potential efficacy of IV and later, SC daclizumab, while continuing to reduce other immunosuppressive medications commensurate with the standard of care. Primary safety outcomes are the discontinuation of study therapy due to reduced vision or the occurrence of adverse events. Secondary outcome measures include visual acuity and the grading of immunosuppressive medications, anterior chamber and vitreous cells, and vitreous haze.

ELIGIBILITY:
* INCLUSION CRITERIA

Participant is 18 years of age or older.

Participant has a diagnosis of sight-threatening, intermediate or posterior uveitis of at least three months duration prior to orginal enrollment, requiring treatment to control their intraocular inflammatory disease with at least 20 mg/day of prednisone (or equivalent) or any combination of two or more anti-inflammatory treatments for uveitis, including for example prednisone, cyclophosphamide, cyclosporine, azathioprine, mycophenolate mofetil, methotrexate, etc.

Participant exhibits intolerance to the indicated systemic medications required for their uveitis or, though their uveitis may be under control, wish to be taken off their present medications due to potential or actual unacceptable side effects.

Participant has visual acuity in at least one eye of 20/63 or better (ETDRS, logMAR less than 0.54).

Participant has normal renal or liver function or evidence of no worse than mild abnormalities as defined by the WHO/NEI criteria.

Participant is not currently pregnant or lactating.

Participant with reproductive potential and who is sexually active agrees to use acceptable birth control methods throughout the course of the study.

EXCLUSION CRITERIA

Participants under the age of 18 years.

Participants who had received previous treatment with an IL-2 directed monoclonal antibody or any other investigational agent that would interfere with the ability to evaluate the safety, efficacy or pharmacokinetics of daclizumab.

Participants with a history or diagnosis of Behcet's disease.

Participant has a significant active infection.

Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past 5 years.

Participant is hypersensitive to fluorescein dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 1996-06-04; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brown PS Jr, Parenteau GL, Dirbas FM, Garsia RJ, Goldman CK, Bukowski MA, Junghans RP, Queen C, Hakimi J, Benjamin WR, et al. Anti-Tac-H, a humanized antibody to the interleukin 2 receptor, prolongs primate cardiac allograft survival. Proc Natl Acad Sci U S A. 1991 Apr 1;88(7):2663-7. doi: 10.1073/pnas.88.7.2663. PMID 2011577